CLINICAL TRIAL: NCT07193069
Title: Clinical and Biological Signs of Dapagliflozin Overdose in ICU Patients With Metformin Poisoning
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0109_REANIMATION_INTEND
Record Dates: First submitted 2025-06-30; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Drug Overdose; Metformin; Dapagliflozin; Lactic Acidosis; Diabetic Ketoacidosis; Intensive Care Units
MeSH Terms: conditions — Drug Overdose; Acidosis, Lactic; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at patients admitted to intensive care for drug poisoning involving metformin, a common diabetes medication. Researchers will compare two groups: patients who overdosed on metformin alone and those who took both metformin and dapagliflozin, another diabetes drug. The goal is to find clinical or laboratory signs that could help doctors quickly recognize a dapagliflozin overdose in this context, which could improve treatment and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Admission to an intensive care unit (ICU) due to acute drug poisoning
* Documented exposure to either:
* Metformin alone
* Metformin in combination with dapagliflozin

Exclusion Criteria:

* Patients under 18 years of age
* No exposure to metformin
* Exposure to dapagliflozin without metformin

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18 years and older) who were admitted to intensive care units across multiple centers for acute drug poisoning involving metformin, with or without dapagliflozin. Participants will be identified retrospectively through case collection from the SRLF (Société de Réanimation de Langue Française) and existing hospital records over the past 10 years. The study will include both cases of isolated metformin overdose and cases of combined metformin and dapagliflozin overdose.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Identification of clinical and biological differences between patients admitted to intensive care for metformin overdose alone versus those with combined metformin and dapagliflozin overdose. | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France